CLINICAL TRIAL: NCT03359577
Title: Randomized, Double Blind, Placebo Controlled Clinical Study to Investigate Efficacy of Psorax35 for Treatment of Psoriasis
Brief Title: Clinical Study to Investigate Psorax35 Supplementation in Patients With Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arctic Nutrition AS (Industry)
Collaborators: University of Bergen (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Psorax35-H17
Record Dates: First submitted 2017-11-15; First posted 2017-12-02 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Chronic plaque psoriasis; Inflammation; Cardiovascular diseases
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psorax35 (Experimental): Food supplement Psorax35 capsules containing fish roe extract high in eicosapentaenoic acid (EPA)/docosahexaenoic acid (DHA) phospholipid. Dose: 10 capsules of 590 mg. Route of administration: oral.
  Interventions: Dietary Supplement: Psorax35
- MCT oil (Placebo Comparator): Placebo capsules containing coconut oil high in caprylic acid C8:0 and capric acid C10:0 (Medium Chain triglycerides (MCT) oil). Dose: 10 capsules of 590 mg: Route of administration: oral.
  Interventions: Dietary Supplement: MCT oil

INTERVENTIONS:
Dietary Supplement: Psorax35 — This is a randomized, 32 weeks, single center, placebo controlled, double blind study to investigate Psorax35 supplementation in patients with mild to moderate Psoriasis. Groups of patients will be block randomized using randomly selected block sizes, and stratified according to gender.
  Arms: Psorax35
Dietary Supplement: MCT oil — This is a randomized, 32 weeks, single center, placebo controlled, double blind study to investigate Psorax35 supplementation in patients with mild to moderate Psoriasis. Groups of patients will be block randomized using randomly selected block sizes, and stratified according to gender.
  Arms: MCT oil

SUMMARY:
The main objective of this study is to establish the efficacy and safety of Psorax35 supplementation in patients with mild to moderate Psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a common, genetically predisposed, inflammatory and proliferative disease of the skin, the most characteristic lesions consisting of chronic, sharply demarcated, dull-red scaly plaques, particularly on extensor parts of limbs and in the scalp. Psoriasis can be divided into mild, moderate or severe psoriasis based on the extent of the skin changes

Psorax35, which is extracted from herring roe are shown to improve the condition of people with psoriasis.

The objective of this study is to investigate the effect, safety, and mechanism of action of Psorax35 on mild to moderate Psoriasis and comorbidities associated with psoriasis through a 32-weeks study.

The participants will be randomized into one of two arms; Psorax35 and Placebo. The study will include a total of 6 treatment visits involving Blood samples, Photo documentation, Psoriasis and Severity index (PASI), Body surface area (BSA), Physician's Static Global Assessment (PSGA), Life quality index (EQ-5D, VAS and DLQI), Blood pressure, Blood rate, Body Mass Index (BMI), Waist circumference, Waist/hip ratio, and 24 hrs dietary recall. At visit 4 Blood samples, Blood pressure, Blood rate, BMI, Waist circumference, Waist/hip ratio, and 24 hrs dietary recall are not included.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male subjects at least 18 years old understanding Norwegian oral and written information
2. Diagnosis of mild to moderate psoriasis vulgaris for at least 6 months prior to mild to moderate Psoriasis vulgaris as defined at screening by:

   * PASI scores less than 10 (mild psoriasis) and
   * Body surface area affected by chronic plaque psoriasis 1%-9.9% (mild and moderate psoriasis)
3. Women of childbearing potential must have a negative serum pregnancy test at the screening visit.

Exclusion Criteria:

1. Pregnancy
2. Initiation of a drug known to cause or exacerbate psoriasis
3. Having received an investigational medical product (IMP) or investigational device within 28 days' prior randomization
4. Alcohol and drug abuse or any condition associated with poor compliance
5. Malabsorption disorder
6. Scheduled hospitalization during the course of the study that could compromise the study
7. Major diseases or infections
8. Known or suspected sensitivity or allergic reactions to the IMP or excipients
9. Presence of other major medical or psychiatric illness that would affect the ability to participate in the study or put the subject at increased risk
10. Planned trip abroad to a sunny resort involving active sun exposure
11. Any anti psoriatic treatment
12. Immunosuppressive - immunomodulating treatment given for any other reason than psoriasis
13. UV treatment and return from a sunny resort involving active sun exposure for the last 4-6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Change in PASI | Baseline to 32 weeks
  Change from baseline in PASI in the Psorax35 group as compared to Placebo at week 32.

SECONDARY OUTCOMES:
Change in PASI over 24 weeks | Baseline to 24 weeks
  Change from baseline in PASI in the Psorax35 group as compared to Placebo at week 6, 12, 18, and 24.
Number of patients achieving PASI<3 | Baseline to 32 weeks
  Number of patients achieving PASI<3 in the Psorax35 group as compared to Placebo at week 6, 12, 18, 24, and 32.
Improvement in PASI | Baseline to 32 weeks
  Difference in 50% improvement in PASI (PASI-50), difference in 75% improvement in PASI (PASI-75) and difference in 90% improvement in PASI (PASI-90) from baseline in the Psorax35 group as compared with Placebo group at week 6, 12, 18, 24, and 32.
Change in Physician's Static Global Assessment (PSGA) | Baseline to 32 weeks
  Changes from baseline in PSGA=0-1 demonstrating clear or almost clear skin in the Psorax35 group as compared to Placebo group at week 6, 12, 18, 24, and 32.
Change in Dermatology Life Quality Index (DLQI) | Baseline to 32 weeks
  Changes from baseline in DLQ index in the Psorax35 group as compared to Placebo at week 6, 12, 18, 24, and 32.
Change in EuroQoL 5 index (EQ-5D) | Baseline to 32 weeks
  Change from baseline in EuroQoL 5 index in the Psorax35 group as compared to Placebo group at week 6, 12, 18, 24, and 32.
Change in Visual analogue scale (VAS) score | Baseline to 32 weeks
  Changes from baseline in VAS Scores (pruritus, pain skin/joints, stinging and total health condition (general/skin)) in the Psorax35 group as compared to Placebo at week 6, 12, 18, 24, and 32.
Changes in highly sensitive C-reactive protein | Baseline to 32 weeks
  Changes from baseline in highly sensitive C-reactive protein (mg/L) in the Psorax35 group as compared to Placebo at week 12, and 32.
Adverse Events (AE) and Severe Adverse Events (SAE) | Baseline to week 32
  Monitoring of AEs and SAEs.
Changes in fasting serum lipids | Baseline to 32 weeks
  Changes from baseline in serum lipids (Triacylglycerol (TAG), total cholesterol (TK), HDL-cholesterol, LDL-cholesterol, free-cholesterol, phospholipids, non-esterified fatty acids, non-HDL-cholesterol - mmol/L) and lipid ratios (TAG/TK ratio, HDL-chol/LDL-chol ratio), in the Psorax35 group as compared to Placebo at week 6, 12, 24, and 32.
Changes in fasting serum glucose | Baseline to 32 weeks
  Changes from baseline in serum glucose (mmol/L) in the Psorax35 group as compared to Placebo at week 6, 12, 24, and 32
Changes in fasting serum insulin and insulin C-peptide | Baseline to 32 weeks
  Changes from baseline in serum insulin (mIE/L) and insulin C-peptide (nmol/L) in the Psorax35 group as compared to Placebo at week 12, and 32.
Changes in fasting serum HbA1c | Baseline to 32 weeks
  Changes from baseline in serum HbA1c (%) in the Psorax35 group as compared to Placebo at week 12, and 32.
Changes in blood pressure | Baseline to 32 weeks
  Changes from baseline in blood pressure (mmHg) in the Psorax35 group as compared to Placebo at week 6, 12, 24, and 32.
Changes in heart rate | Baseline to 32 weeks
  Changes from baseline in heart rate (bpm) in the Psorax35 group as compared to Placebo at week 6, 12, 24, and 32.
Changes in Body Mass Index (BMI) | Baseline to 32 weeks
  Changes from baseline in Body Mass Index (BMI) in the Psorax35 group as compared to Placebo at week 6, 12, 24, and 32.
  Weight in kilograms and height in meters will be combined to report BMI in kg/m2
Changes in waist/hip ratio | Baseline to 32 weeks
  Changes from baseline in waist/hip ratio in the Psorax35 group as compared to Placebo at week 6, 12, 24, and 32.
  Waist in centimeters and hip in centimeters will be combined to report waist/hip ratio.
Changes in plasma cytokines including adipocytokines | Baseline to 32 weeks
  Changes from baseline in plasma cytokines including adipocytokines (pg/mL) in the Psorax35 group as compared to Placebo group at week 12, and 32.
Changes in serum antioxidant capacity | Baseline to 32 weeks
  Changes from baseline in serum antioxidant capacity (nmol Trolox ekv./ul) in the Psorax35 group as compared to Placebo group at week 12, and 32.
Changes in serum Vitamin D | Baseline to 32 weeks
  Changes from baseline in serum Vitamin D (nmol/L) in the psorax35 group as compared to Placebo group at week 12, and 32.
Difference in use of cream-based treatment | Baseline to 32 weeks
  Difference in use of rescue medication from baseline in the Psorax35 group as compared to placebo group at week 6, 12, 18, 24, and 32.
  Amount of cream-based treatment in grams and number of days treated will be combined to report the use.
Changes in safety laboratory parameters including hematology, clinical chemistry | Baseline to 32 weeks
  Changes from baseline in safety laboratory parameters including hematology (Hemoglobin-g/dL, Hematocrit, Erythrocytes-10^9/L, Leukocytes-10^9/L, Lymphocytes-10^9/L, Monocytes-10^9/L, Eosinophiles-10^9/L, Neutrophiles-10^9/L, Blood plates-10^9/L), and clinical chemistry (ALAT-u/L, lactate dehydrogenase-u/L, creatine kinase-u/L, creatinine-umol/L, gamma-glutamyltransferase-u/L).

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Berge, PhD, Principal Investigator — University of Bergen
Locations (1):
- Haukeland Universitetssjukehus, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tveit KS, Brokstad KA, Berge RK, Saebo PC, Hallaraker H, Brekke S, Meland N, Bjorndal B. A Randomized, Double-blind, Placebo-controlled Clinical Study to Investigate the efficacy of Herring Roe Oil for treatment of Psoriasis. Acta Derm Venereol. 2020 May 28;100(10):adv00154. doi: 10.2340/00015555-3507. PMID 32378724